CLINICAL TRIAL: NCT04661839
Title: A Phase 1, Double-blind, Randomized, Placebo-controlled Study to Evaluate Safety and Pharmacokinetics of Anti-SARS-CoV-2 Immunoglobulin Intravenous (Human) Investigational Product (COVID-HIGIV) Administered as a Single Dose Regimen to Healthy Adults
Brief Title: A COVID-19 Study to Evaluate Safety and Pharmacokinetics of COVID-HIGIV Administered in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EBS-CVH-003
Record Dates: First submitted 2020-12-09; First posted 2020-12-10 (Actual); Results first posted 2023-02-02 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Coronavirus disease 2019; Severe acute respiratory syndrome coronavirus 2; Immunoglobulins; Immunoglobulins, Intravenous; Antibodies
MeSH Terms: conditions — COVID-19 | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- COVID-HIGIV Dose Level 1 (100 mg/kg) (Experimental): Eligible subjects randomized to receive a single IV infusion of COVID-HIGIV dose level 1 (100 mg/kg).
  Interventions: Biological: COVID-HIGIV
- COVID-HIGIV Dose Level 2 (200 mg/kg) (Experimental): Eligible subjects randomized to receive a single IV infusion of COVID-HIGIV dose level 2 (200 mg/kg).
  Interventions: Biological: COVID-HIGIV
- COVID-HIGIV Dose Level 3 (400 mg/kg) (Experimental): Eligible subjects randomized to receive a single IV infusion of COVID-HIGIV dose level 3 (400 mg/kg).
  Interventions: Biological: COVID-HIGIV
- Dose Placebo (saline) (Placebo Comparator): Eligible subjects randomized to receive a single IV infusion of saline placebo.
  Interventions: Other: Placebo (saline)

INTERVENTIONS:
Biological: COVID-HIGIV — COVID-HIGIV is a purified immunoglobulin G (IgG) liquid preparation containing antibodies (including neutralizing antibodies) to SARS-CoV-2. COVID-HIGIV will be administered via intravenous infusion.
  Other Names: NP-028
  Arms: COVID-HIGIV Dose Level 1 (100 mg/kg); COVID-HIGIV Dose Level 2 (200 mg/kg); COVID-HIGIV Dose Level 3 (400 mg/kg)
Other: Placebo (saline) — The reference product is a liquid solution of normal saline (0.9% weight per unit volume (w/v) sodium chloride). Placebo will be administered via intravenous infusion.
  Arms: Dose Placebo (saline)

SUMMARY:
This study is designed to evaluate three dose levels of Anti-SARS-CoV-2 Immunoglobulin Intravenous (Human) (COVID-HIGIV) for safety and pharmacokinetics (PK) in healthy adults. Twenty-eight healthy adult subjects will be enrolled into the study to receive a single dose of COVID-HIGIV or placebo with 84 days of safety and PK follow-up post-administration.

DETAILED DESCRIPTION:
This study will be a Phase 1, single-center, randomized, double-blind, placebo-controlled design to assess safety and PK of COVID-HIGIV in healthy adults.

In total, 28 healthy adult subjects are to be enrolled and randomized 2:2:2:1 into four study treatment arms to receive a single intravenous (IV) infusion of one of three COVID-HIGIV dose levels or saline placebo, respectively.

The enrollment/dosing of the first seven subjects in the study will be staggered. Available safety data will be reviewed by Study Monitoring Committee (SMC) after seven subjects have completed at least 72 hours of safety follow-up. Subjects will be followed up for safety and PK up to 84 days post-administration.

The SMC will perform overall ongoing review of safety data during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent (voluntarily signed by the subject) prior to performing study procedures.
2. Females and males 18-60 years of age, inclusive.
3. Have a body mass index (BMI) less than or equal to 35.0 kg/m2.
4. Women who are either:

   A) Not of childbearing potential: either surgically sterile (at least six weeks post bilateral tubal ligation, bilateral oophorectomy or hysterectomy); or post-menopausal (defined as ≥50 years of age with a history of ≥12 months without menses prior to randomization in the absence of other pathologic or physiologic causes, following cessation of exogenous sex-hormonal treatment); OR

   B) Women of childbearing potential (WOCBP) who are not planning to be pregnant during the study period and meet all of the following criteria:

   Negative serum pregnancy test (PT) at Screening; and Negative PT prior to dosing at Day 1; and

   Use of a highly effective contraception during the study period:
   * Hormonal contraceptives (e.g., implants, pills, patches) initiated ≥30 days prior to Day 1; or
   * Intrauterine device (IUD) inserted ≥30 days prior to Day 1; or
   * Double barrier type of birth control (e.g., male condom with female diaphragm, male condom with cervical cap).
5. Subject understands and agrees to comply with planned study procedures.
6. Healthy as determined by the Principal Investigator based on medical history, physical exam, vital signs, urinalysis, blood chemistry and hematology test results at Screening and evidence of no prior exposure to SARS-CoV-2 (i.e., Reverse transcription polymerase chain reaction [RT-PCR] negative for SARS-CoV-2 and negative for SARS-CoV-2 antibodies) at Screening.

Exclusion Criteria:

1. Use of any investigational product, within 30 days prior to Screening, or use of investigational SARS-CoV-2 vaccines, SARS-CoV-2 monoclonal antibodies or COVID-19 convalescent plasma at any time prior to Screening or during the study follow-up period, or subject plans to participate in another clinical study during the study period.
2. Screening clinical laboratory test result greater than the laboratory's upper limit of normal (ULN) for alanine aminotransferase (ALT), aspartate aminotransferase (AST), random glucose, total and/or bilirubin, blood urea nitrogen (BUN), or creatinine. Other serum chemistry parameters that are not within the reference range will not be considered exclusionary unless deemed clinically significant by the Principal Investigator.
3. History of allergy or hypersensitivity to blood or plasma products or to COVID-HIGIV excipients (proline, PS80).
4. History of allergy to latex or rubber.
5. History of hemolytic anemia.
6. History of Immunoglobulin A (IgA) deficiency.
7. Receipt of any blood product within the past 12 months.
8. Plasma donation within 7 days or significant blood loss or blood donation within 56 days of randomization/dosing.
9. History of known congenital or acquired immunodeficiency or receipt of immunosuppressive therapy (e.g., prednisone or equivalent for more than two consecutive weeks within the past three months).
10. History of thrombosis or hypercoagulable state with increased risk of thrombosis.
11. History of clinically significant chronic illness (e.g., requiring hospitalization in the past three months) such as cardiac, pulmonary, renal, hepatic or other chronic conditions.
12. Receipt of a live vaccine within 28 days prior to screening or anticipated receipt of a live vaccine during the study period.
13. Currently pregnant, breastfeeding, or planning to become pregnant during the study.
14. History of, or suspected substance abuse problem (including alcohol).
15. Other medical condition which may place subject at increased risk due to participation in the study as determined by the investigator.
16. Any planned elective surgery during the study period.
17. An opinion of the investigator that it would be unwise to allow the individual to be randomized into the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2020-12-24 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Cabell, MD, MHS, Study Director — Emergent BioSolutions
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and Statistical Analysis Plan (redacted) to be shared.
Supporting Information: Study Protocol, SAP
Time Frame: By April 2025 for up to 2 years

REFERENCES:
- [Derived] Liu STH, Mirceta M, Lin G, Anderson DM, Broomes T, Jen A, Abid A, Reich D, Hall C, Aberg JA. Safety, Tolerability, and Pharmacokinetics of Anti-SARS-CoV-2 Immunoglobulin Intravenous (Human) Investigational Product (COVID-HIGIV) in Healthy Adults: a Randomized, Controlled, Double-Blinded, Phase 1 Study. Antimicrob Agents Chemother. 2023 Mar 16;67(3):e0151422. doi: 10.1128/aac.01514-22. Epub 2023 Feb 28. PMID 36852998

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | COVID-HIGIV Dose Level 1 (100 mg/kg) | COVID-HIGIV Dose Level 2 (200 mg/kg) | COVID-HIGIV Dose Level 3 (400 mg/kg) | Dose Placebo (Saline)
Started | 8 | 8 | 8 | 4
Safety Population | 8 | 8 | 7 | 4
Completed | 7 | 8 | 7 | 3
Not Completed | 1 | 0 | 1 | 1
Not completed — Not Treated | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Data is from the safety population which includes all subjects who received any amount of study treatment.
Groups:
- COVID-HIGIV Dose Level 1 (100 mg/kg): Eligible subjects will be randomized to receive a single IV infusion of COVID-HIGIV dose level 1 (100 mg/kg).
  COVID-HIGIV: COVID-HIGIV is a purified immunoglobulin G (IgG) liquid preparation containing antibodies (including neutralizing antibodies) to SARS-CoV-2. COVID-HIGIV will be administered via intravenous infusion.
- COVID-HIGIV Dose Level 2 (200 mg/kg): Eligible subjects will be randomized to receive a single IV infusion of COVID-HIGIV dose level 2 (200 mg/kg).
  COVID-HIGIV: COVID-HIGIV is a purified immunoglobulin G (IgG) liquid preparation containing antibodies (including neutralizing antibodies) to SARS-CoV-2. COVID-HIGIV will be administered via intravenous infusion.
- COVID-HIGIV Dose Level 3 (400 mg/kg): Eligible subjects will be randomized to receive a single IV infusion of COVID-HIGIV dose level 3 (400 mg/kg).
  COVID-HIGIV: COVID-HIGIV is a purified immunoglobulin G (IgG) liquid preparation containing antibodies (including neutralizing antibodies) to SARS-CoV-2. COVID-HIGIV will be administered via intravenous infusion.
- Dose Placebo (Saline): Eligible subjects will be randomized to receive a single IV infusion of saline placebo.
  Placebo (saline): The reference product is a liquid solution of normal saline (0.9% weight per unit volume (w/v) sodium chloride). Placebo will be administered via intravenous infusion.
- Total: Total of all reporting groups
Arm/Group | COVID-HIGIV Dose Level 1 (100 mg/kg) | COVID-HIGIV Dose Level 2 (200 mg/kg) | COVID-HIGIV Dose Level 3 (400 mg/kg) | Dose Placebo (Saline) | Total
Number analyzed (Participants) | 8 | 8 | 7 | 4 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.4 (10.2) | 31.5 (9.5) | 33.9 (14.0) | 27.8 (8.3) | 30.6 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 1 | 10
  Male | 5 | 5 | 4 | 3 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3 | 2 | 8
  Not Hispanic or Latino | 7 | 6 | 4 | 2 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 1 | 7
  White | 5 | 5 | 3 | 1 | 14
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 2 | 2 | 5
Height [Mean (Standard Deviation); unit: centimeters] | 173.0 (8.9) | 172.1 (12.2) | 168.4 (12.3) | 184.8 (14.9) | 173.3 (12.2)
Baseline weight [Mean (Standard Deviation); unit: kilograms] | 72.2 (11.9) | 79.3 (12.4) | 74.1 (15.9) | 80.8 (15.7) | 76.1 (13.4)
Baseline body mass index [Mean (Standard Deviation); unit: kilograms per meter squared (kg/m^2)] | 24.1 (3.7) | 26.9 (4.5) | 25.9 (3.2) | 23.5 (1.2) | 25.3 (3.7)

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Adverse Events (AEs) up to 3 Days Post-dosing
Description: Number of subjects with AEs and severity of AEs up to 3 days post-dosing.
Time Frame: Day 1 through Day 4
Population: Safety population includes all subjects who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-HIGIV Dose Level 1 (100 mg/kg) | COVID-HIGIV Dose Level 2 (200 mg/kg) | COVID-HIGIV Dose Level 3 (400 mg/kg) | Dose Placebo (Saline)
Number analyzed (Participants) | 8 | 8 | 7 | 4
Participants
  Subjects with an adverse event (AE) | 3 | 4 | 6 | 2
  Subjects with a severe adverse event (SAE) | 0 | 0 | 0 | 0

2. Primary Outcome: Subjects With Adverse Events That Led to Discontinuation or Temporary Suspension of IV Infusion
Description: Number of subjects and severity of treatment emergent adverse events (TEAEs) that led to discontinuation or temporary suspension of IV infusion.
Time Frame: 0 hours to 2.5 hours
Population: Safety population includes all subjects who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-HIGIV Dose Level 1 (100 mg/kg) | COVID-HIGIV Dose Level 2 (200 mg/kg) | COVID-HIGIV Dose Level 3 (400 mg/kg) | Dose Placebo (Saline)
Number analyzed (Participants) | 8 | 8 | 7 | 4
Participants
  Any TEAE leading to infusion interruption | 1 | 1 | 1 | 0
  Any TEAE leading to infusion discontinuation | 0 | 0 | 0 | 0

3. Primary Outcome: Subjects With AEs and SAEs After IV Infusion
Description: Number of subjects with TEAEs and SAEs up to 84 days post-dosing.
Time Frame: Day 1 through Day 85
Population: Safety population includes all subjects who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-HIGIV Dose Level 1 (100 mg/kg) | COVID-HIGIV Dose Level 2 (200 mg/kg) | COVID-HIGIV Dose Level 3 (400 mg/kg) | Dose Placebo (Saline)
Number analyzed (Participants) | 8 | 8 | 7 | 4
Participants
  Number of subjects with any TEAE | 3 | 6 | 6 | 3
  Number of subjects with serious adverse events (SAEs) | 0 | 0 | 0 | 1

4. Primary Outcome: Total Number of AEs and SAEs After IV Infusion
Description: Number of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) in all subjects reporting TEAEs/SAEs up to 84 days post-dosing.
Time Frame: Day 1 through Day 85
Population: Safety population includes all subjects who received any amount of study treatment.
Measure: Number; unit: Events
Arm/Group | COVID-HIGIV Dose Level 1 (100 mg/kg) | COVID-HIGIV Dose Level 2 (200 mg/kg) | COVID-HIGIV Dose Level 3 (400 mg/kg) | Dose Placebo (Saline)
Number analyzed (Participants) | 8 | 8 | 7 | 4
Events
  Total number of adverse events (AEs) for all subjects reporting TEAEs | 5 | 18 | 19 | 8
  Total number of SAEs for all subjects reporting SAEs | 0 | 0 | 0 | 1

5. Primary Outcome: Pharmacokinetics (PK) Parameter of Area Under the Concentration-time Curve (AUC) From Time 0 to the Last Quantifiable Concentration (AUC0-last) of SARS-CoV-2 Antibodies After Dose of COVID-HIGIV
Description: The area under the concentration-time curve from time 0 to the last quantifiable concentration of SARS-CoV-2 binding IgG antibodies after COVID-HIGIV dose. Data for PK calculations was collected: pre-dose within 2 hrs prior to dosing, and post-dose at: 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, Day 4, Day 8, Day 15, Day 22, Day 29, Day 43, Day 57 and Day 85.
Time Frame: Day 1 through Day 85
Population: The PK population included all subjects who received COVID-HIGIV and had an adequate set of evaluable PK samples (a suitable predose sample and at least one measurable postdose sample).
Measure: Geometric Mean (95% Confidence Interval); unit: h*Alliance Units (AU)/mL
Arm/Group | COVID-HIGIV Dose Level 1 (100 mg/kg) | COVID-HIGIV Dose Level 2 (200 mg/kg) | COVID-HIGIV Dose Level 3 (400 mg/kg)
Number analyzed (Participants) | 7 | 8 | 7
h*Alliance Units (AU)/mL | 2961.93 [2246.17 to 3905.77] | 6678.80 [6014.80 to 7416.11] | 11722.82 [10108.67 to 13594.72]

6. Primary Outcome: Pharmacokinetics Parameter of Area Under the Concentration-time (AUC) From Time 0 to Infinity (AUC0-inf) After Dose of COVID-HIGIV
Description: Area under the concentration-time curve from time 0 to the last quantifiable concentration plus the additional area extrapolated to infinity of SARS-CoV-2 binding IgG antibodies after COVID-HIGIV dose. Data for PK calculations was collected: pre-dose within 2 hrs prior to dosing, and post-dose at: 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, Day 4, Day 8, Day 15, Day 22, Day 29, Day 43, Day 57 and Day 85.
Time Frame: Day 1 through Day 85
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: h*AU/mL
Arm/Group | COVID-HIGIV Dose Level 1 (100 mg/kg) | COVID-HIGIV Dose Level 2 (200 mg/kg) | COVID-HIGIV Dose Level 3 (400 mg/kg)
Number analyzed (Participants) | 6 | 8 | 7
h*AU/mL | 3818.25 [2729.49 to 5341.31] | 8255.74 [7341.21 to 9284.19] | 13028.08 [11014.89 to 15409.22]

7. Primary Outcome: Pharmacokinetics Parameter of Area Under the Concentration-time Curve (AUC) From Time 0 to 14 Days After Dose of COVID-HIGIV
Description: AUC from time 0 to 14 days (AUC0-14d) of SARS-CoV-2 binding IgG antibodies after COVID-HIGIV. Data for PK calculations was collected: pre-dose within 2 hrs prior to dosing, and post-dose at: 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, Day 4, Day 8, and Day 15.
Time Frame: Day 1 through Day 15
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: h*AU/mL
Arm/Group | COVID-HIGIV Dose Level 1 (100 mg/kg) | COVID-HIGIV Dose Level 2 (200 mg/kg) | COVID-HIGIV Dose Level 3 (400 mg/kg)
Number analyzed (Participants) | 5 | 7 | 7
h*AU/mL | 3398.55 [2579.60 to 4477.49] | 6834.66 [6142.30 to 7605.06] | 11722.82 [10108.67 to 13594.72]

8. Primary Outcome: Pharmacokinetics Parameter of Area Under the Concentration-time Curve (AUC) From Time 0 to 28 Days (AUC0-28d) After Dose of COVID-HIGIV
Description: AUC from time 0 to 28 days of SARS-CoV-2 binding IgG antibodies after COVID-HIGIV dose. Data for PK calculations was collected: pre-dose within 2 hrs prior to dosing, and post-dose at: 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, Day 4, Day 8, Day 15, Day 22, and Day 29.
Time Frame: Day 1 through Day 29
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: h*AU/mL
Arm/Group | COVID-HIGIV Dose Level 1 (100 mg/kg) | COVID-HIGIV Dose Level 2 (200 mg/kg) | COVID-HIGIV Dose Level 3 (400 mg/kg)
Number analyzed (Participants) | 7 | 8 | 6
h*AU/mL | 2961.93 [2246.17 to 3905.77] | 6678.80 [6014.80 to 7416.11] | 11296.33 [9765.56 to 13067.06]

9. Primary Outcome: Pharmacokinetics Parameter of Maximum Observed Concentration (Cmax) of SARS-CoV-2 Antibodies Observed After Dose of COVID-HIGIV
Description: The Cmax of SARS-CoV-2 binding IgG antibodies observed after COVID-HIGIV dose. Data for PK calculations was collected: pre-dose within 2 hrs prior to dosing, and post-dose at: 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, Day 4, Day 8, Day 15, Day 22, Day 29, Day 43, Day 57 and Day 85.
Time Frame: Day 1 through Day 85
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | COVID-HIGIV Dose Level 1 (100 mg/kg) | COVID-HIGIV Dose Level 2 (200 mg/kg) | COVID-HIGIV Dose Level 3 (400 mg/kg)
Number analyzed (Participants) | 7 | 8 | 7
AU/mL | 7.69 [6.60 to 8.97] | 17.02 [15.63 to 18.54] | 33.27 [28.69 to 38.58]

10. Primary Outcome: Pharmacokinetics Parameter of Time at Which Cmax Occurs After Dose of COVID-HIGIV
Description: Time at which Cmax occurs (Tmax) after COVID-HIGIV at each dose level .Data for PK calculations was collected: pre-dose within 2 hrs prior to dosing, and post-dose at: 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, Day 4, Day 8, Day 15, Day 22, Day 29, Day 43, Day 57 and Day 85.
Time Frame: Day 1 through Day 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | COVID-HIGIV Dose Level 1 (100 mg/kg) | COVID-HIGIV Dose Level 2 (200 mg/kg) | COVID-HIGIV Dose Level 3 (400 mg/kg)
Number analyzed (Participants) | 7 | 8 | 7
hours | 7.09 (7.84) | 7.93 (6.81) | 5.36 (1.46)

11. Primary Outcome: Pharmacokinetics Parameter of Trough Concentration of SARS-CoV-2 Antibodies Observed 28 Days After Dose (Cmin28d) of COVID-HIGIV
Description: The observed trough concentration of SARS-CoV-2 binding IgG antibodies 28 days after COVID-HIGIV dose. Data for PK calculations was collected: pre-dose within 2 hrs prior to dosing, and post-dose at: 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, Day 4, Day 8, Day 15, Day 22, and Day 29.
Time Frame: Day 1 through Day 29
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | COVID-HIGIV Dose Level 1 (100 mg/kg) | COVID-HIGIV Dose Level 2 (200 mg/kg) | COVID-HIGIV Dose Level 3 (400 mg/kg)
Number analyzed (Participants) | 7 | 8 | 6
AU/mL | 2.06 [1.31 to 3.22] | 3.33 [2.99 to 3.70] | 5.47 [4.56 to 6.56]

12. Primary Outcome: Pharmacokinetics Parameter of Apparent Terminal Elimination Half-life (T1/2) After Dose of COVID-HIGIV
Description: The apparent terminal elimination half-life (T1/2) after dose of COVID-HIGIV. Data for PK calculations was collected: pre-dose within 2 hrs prior to dosing, and post-dose at: 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, Day 4, Day 8, Day 15, Day 22, Day 29, Day 43, Day 57 and Day 85.
Time Frame: Day 1 through Day 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | COVID-HIGIV Dose Level 1 (100 mg/kg) | COVID-HIGIV Dose Level 2 (200 mg/kg) | COVID-HIGIV Dose Level 3 (400 mg/kg)
Number analyzed (Participants) | 6 | 8 | 7
hours | 583.13 (237.39) | 752.87 (257.67) | 618.79 (148.64)

13. Primary Outcome: Pharmacokinetics Parameter of Systemic Clearance (CL) After Dose of COVID-HIGIV
Description: The systemic clearance (CL) of SARS-CoV-2 binding IgG antibodies after dose of COVID-HIGIV. Data for PK calculations was collected: pre-dose within 2 hrs prior to dosing, and post-dose at: 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, Day 4, Day 8, Day 15, Day 22, Day 29, Day 43, Day 57 and Day 85.
Time Frame: Day 1 through Day 85
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: mL/h
Arm/Group | COVID-HIGIV Dose Level 1 (100 mg/kg) | COVID-HIGIV Dose Level 2 (200 mg/kg) | COVID-HIGIV Dose Level 3 (400 mg/kg)
Number analyzed (Participants) | 6 | 8 | 7
mL/h | 0.0194 [0.0138 to 0.0272] | 0.0188 [0.0156 to 0.0227] | 0.0223 [0.0176 to 0.0284]

14. Primary Outcome: Pharmacokinetics Parameter of Volume of Distribution (Vz) After Dose of COVID-HIGIV
Description: The volume of distribution (Vz) of SARS-CoV-2 binding IgG antibodies after dose of COVID-HIGIV. Data for PK calculations was collected: pre-dose within 2 hrs prior to dosing, and post-dose at: 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, Day 4, Day 8, Day 15, Day 22, Day 29, Day 43, Day 57 and Day 85.
Time Frame: Day 1 through Day 85
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: mL
Arm/Group | COVID-HIGIV Dose Level 1 (100 mg/kg) | COVID-HIGIV Dose Level 2 (200 mg/kg) | COVID-HIGIV Dose Level 3 (400 mg/kg)
Number analyzed (Participants) | 6 | 8 | 7
mL | 15.19 [11.74 to 19.65] | 19.72 [17.01 to 22.86] | 19.40 [16.20 to 23.23]

15. Secondary Outcome: Body-weight Normalized Pharmacokinetics Parameter of Maximum Observed Concentration of SARS-CoV-2 Antibodies Observed After Dose of COVID-HIGIV
Description: The body-weight normalized Cmax (CmaxBWN) of SARS-CoV-2 binding antibodies observed after COVID-HIGIV dose. Data for PK calculations was collected: pre-dose within 2 hrs prior to dosing, and post-dose at: 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, Day 4, Day 8, Day 15, Day 22, Day 29, Day 43, Day 57 and Day 85.
Time Frame: Day 1 through Day 85
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL/kg
Arm/Group | COVID-HIGIV Dose Level 1 (100 mg/kg) | COVID-HIGIV Dose Level 2 (200 mg/kg) | COVID-HIGIV Dose Level 3 (400 mg/kg)
Number analyzed (Participants) | 7 | 8 | 7
AU/mL/kg | 0.11 [0.09 to 0.14] | 0.22 [0.19 to 0.26] | 0.45 [0.39 to 0.53]

16. Secondary Outcome: Body-weight Normalized Pharmacokinetics Parameter of Area Under the Concentration-time Curve (AUC) From Time 0 to the Last Quantifiable Concentration (AUC0-last) of SARS-CoV-2 Antibodies After Dose of COVID-HIGIV
Description: The body-weight normalized area under the concentration-time curve from time 0 to the last quantifiable concentration of SARS-CoV-2 binding IgG antibodies after COVID-HIGIV dose. Data for PK calculations was collected: pre-dose within 2 hrs prior to dosing, and post-dose at: 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, Day 4, Day 8, Day 15, Day 22, Day 29, Day 43, Day 57 and Day 85.
Time Frame: Day 1 through Day 85
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: h*AU/mL/kg
Arm/Group | COVID-HIGIV Dose Level 1 (100 mg/kg) | COVID-HIGIV Dose Level 2 (200 mg/kg) | COVID-HIGIV Dose Level 3 (400 mg/kg)
Number analyzed (Participants) | 7 | 8 | 7
h*AU/mL/kg | 41.83 [30.11 to 58.12] | 85.23 [71.82 to 101.14] | 161.44 [129.11 to 201.87]

17. Secondary Outcome: Body-weight Normalized Pharmacokinetics Parameter of Area Under the Concentration-time (AUC) From Time 0 to the Last Quantifiable Concentration of SARS-CoV-2 Antibodies Plus the Additional Area Extrapolated to Infinity (AUC0-inf) After Dose of COVID-HIGIV
Description: The body-weight normalized area under the concentration-time curve from time 0 to the last quantifiable concentration plus the additional area extrapolated to infinity of SARS-CoV-2 binding IgG antibodies after COVID-HIGIV dose. Data for PK calculations was collected: pre-dose within 2 hrs prior to dosing, and post-dose at: 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, Day 4, Day 8, Day 15, Day 22, Day 29, Day 43, Day 57 and Day 85.
Time Frame: Day 1 through Day 85
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: h*AU/mL/kg
Arm/Group | COVID-HIGIV Dose Level 1 (100 mg/kg) | COVID-HIGIV Dose Level 2 (200 mg/kg) | COVID-HIGIV Dose Level 3 (400 mg/kg)
Number analyzed (Participants) | 6 | 8 | 7
h*AU/mL/kg | 52.07 [36.85 to 73.56] | 105.39 [87.53 to 126.89] | 179.39 [139.91 to 230.02]

18. Secondary Outcome: Body-weight Normalized Pharmacokinetics Parameter of Area Under the Concentration-time Curve (AUC) From Time 0 to 14 Days (AUC0-14d) After Dose of COVID-HIGIV
Description: Body-weight normalized AUC from time 0 to 14 days of SARS-CoV-2 binding IgG antibodies after COVID-HIGIV. Data for PK calculations was collected: pre-dose within 2 hrs prior to dosing, and post-dose at: 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, Day 4, Day 8, and Day 15.
Time Frame: Day 1 through Day 15
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: h*AU/mL/kg
Arm/Group | COVID-HIGIV Dose Level 1 (100 mg/kg) | COVID-HIGIV Dose Level 2 (200 mg/kg) | COVID-HIGIV Dose Level 3 (400 mg/kg)
Number analyzed (Participants) | 5 | 7 | 7
h*AU/mL/kg | 45.90 [28.37 to 74.25] | 87.73 [72.74 to 105.82] | 161.44 [129.11 to 201.87]

19. Secondary Outcome: Body-weight Normalized Pharmacokinetics Parameter of Area Under the Concentration-time Curve (AUC) From Time 0 to 28 Days (AUC0-28d) After Dose of COVID-HIGIV
Description: as for outcome 8
Time Frame: Day 1 through Day 29
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: h*AU/mL/kg
Arm/Group | COVID-HIGIV Dose Level 1 (100 mg/kg) | COVID-HIGIV Dose Level 2 (200 mg/kg) | COVID-HIGIV Dose Level 3 (400 mg/kg)
Number analyzed (Participants) | 7 | 8 | 6
h*AU/mL/kg | 41.83 [30.11 to 58.12] | 85.23 [71.82 to 101.14] | 161.17 [122.08 to 212.77]

20. Secondary Outcome: Body-weight Normalized Pharmacokinetics Parameter of Trough Concentration of SARS-CoV-2 Antibodies Observed 28 Days After Dose (Cmin28d) of COVID-HIGIV
Description: The body-weight normalized observed trough concentration of SARS-CoV-2 binding IgG antibodies 28 days after COVID-HIGIV dose. Data for PK calculations was collected: pre-dose within 2 hrs prior to dosing, and post-dose at: 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, Day 4, Day 8, Day 15, Day 22, and Day 29.
Time Frame: Day 1 through Day 29
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL/kg
Arm/Group | COVID-HIGIV Dose Level 1 (100 mg/kg) | COVID-HIGIV Dose Level 2 (200 mg/kg) | COVID-HIGIV Dose Level 3 (400 mg/kg)
Number analyzed (Participants) | 7 | 8 | 6
AU/mL/kg | 0.0291 [0.0172 to 0.0494] | 0.0425 [0.0371 to 0.0487] | 0.0780 [0.0568 to 0.1072]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Day 1 (Dosing Day) through Day 85 or early withdrawal.
Description: Adverse events were unsolicited.
Arm/Group | COVID-HIGIV Dose Level 1 (100 mg/kg) | COVID-HIGIV Dose Level 2 (200 mg/kg) | COVID-HIGIV Dose Level 3 (400 mg/kg) | Dose Placebo (Saline)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/7 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/7 | 1/4
Other Adverse Events (participants affected / at risk) | 3/8 | 6/8 | 6/7 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COVID-HIGIV Dose Level 1 (100 mg/kg) (N=8) | COVID-HIGIV Dose Level 2 (200 mg/kg) (N=8) | COVID-HIGIV Dose Level 3 (400 mg/kg) (N=7) | Dose Placebo (Saline) (N=4)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COVID-HIGIV Dose Level 1 (100 mg/kg) (N=8) | COVID-HIGIV Dose Level 2 (200 mg/kg) (N=8) | COVID-HIGIV Dose Level 3 (400 mg/kg) (N=7) | Dose Placebo (Saline) (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Xerosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 5 (6) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/39/NCT04661839/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT04661839/SAP_001.pdf